CLINICAL TRIAL: NCT06256146
Title: Investigating Modified Protocols of Oral Immunotherapy to Validate Efficacy and Safety
Acronym: IMPROVES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Moshe Ben-Shoshan, Assistant Professor of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-8424
Record Dates: First submitted 2023-07-06; First posted 2024-02-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Peanut Allergy; Milk Allergy, Cow's; Egg Allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Milk Hypersensitivity; Egg Hypersensitivity | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Protocol - High Dose Arm (Experimental): Subjects will progress through desensitization to a high maintenance dose - 1200 mg of crushed peanut, 200 ml of milk or 1200 mg of egg powder.
  Interventions: Other: Food allergy desensitization / Oral Immunotherapy
- Modified Protocol - Low Dose Arm (Experimental): Subjects will progress through desensitization to a low maintenance dose - 120 mg of crushed peanut, 50 ml of milk or 300 mg of egg powder.
  Interventions: Other: Food allergy desensitization / Oral Immunotherapy
- Modified Protocol - Cooked/Transformed Allergen Arm (Experimental): Subjects will begin desensitization with cooked versions of the allergen (muffins in the case of egg and milk) or transformed versions (Bamba puffs for peanut). They will progress up to a full muffin or 4 Bamba puffs (for egg/milk and peanut respectively). Once subjects have reached these doses, they will transition to doses of pure allergen. They will then progress to the same top dose as subjects in the High Dose Arm.
  Interventions: Other: Food allergy desensitization / Oral Immunotherapy

INTERVENTIONS:
Other: Food allergy desensitization / Oral Immunotherapy — Participants consume increasing doses of allergenic food daily until they reach a maintenance dose. In the case of the High Dose Arm, participants will progress to a daily dose of either 1200 mg, 300 mg or 200 ml of egg, peanut or milk respectively.
  Participants randomized to the Low Dose Arm also begin by consuming small amounts of the allergenic food, gradually increasing the daily dose. However, participants in this group only progress to 300 ml, 30 mg or 50 ml daily dose of egg, peanut or milk respectively.
  The Cooked/Transformed Allergen Arm begins the desensitization with a cooked or transformed form of the allergen - muffins in the case of egg or milk, Bamba puffs in the case of peanut. Participants take increasing amounts of these products (one muffin for egg and milk and four Bamba puffs for peanut) then transition to egg, milk or peanut. Participants then continue their dose progression, getting to 1200 mg, 200 ml or 300 mg for egg, milk and peanut respectively.

SUMMARY:
Protocols for Oral Immunotherapy (OIT) for the main food allergens have been recently incorporated in clinical practice for food allergies and their clinical benefits have been acknowledged in European and Canadian official guidelines. There has been some reluctance in both clinicians and patients to implement these therapies, primarily because of the risk of allergic reactions during the desensitization process. This study will investigate if protocols using low doses of a food allergen or processed versions of the allergen can be both effective in conferring desensitization while inducing fewer allergic symptoms during the desensitization process.

ELIGIBILITY:
Inclusion Criteria:

* A history suggestive of immediate allergy to the food. A convincing clinical history of an IgE mediated reaction to a specific food will be defined as a minimum of 2 mild signs/symptoms or 1 moderate or 1 severe sign/symptom that was likely IgE mediated and occurred within 120 minutes after ingestion or contact
* The presence of at least one of the following confirmatory tests:

  * Positive SPT to the culprit food allergen (weal diameter 3 mm larger than that of the normal saline control). The allergens used will be commercial extracts of the foods (Omega Labs, Toronto, Ontario).
  * Detection of serum specific IgE (>0.35 kU/L) to the culprit food or any of its proteins, measured by fluorescence enzyme immunoassay (Phadia, CAP System, Uppsala, Sweden).

Exclusion Criteria:

* Patients who have uncontrolled respiratory disease (asthma, cystic fibrosis, etc.)
* Patients who present with intercurrent disease active at the time of starting desensitization.
* Non IgE mediated or non-immunological adverse reactions to milk or peanuts.
* Malignant or immunopathological diseases and/or severe primary or secondary immune deficiencies.
* Patients receiving oral immunosuppressor therapy.
* Patients receiving β-blockers (including topical formulations), or who receive daily doses of NSAIDs, aspirin or ACE inhibitors for cardiac issues.
* Associated diseases contraindicating the use of epinephrine: cardiovascular disease, severe hypertension or hypotension.
* Patients diagnosed with eosinophilic gastrointestinal disorders, including patients with a history of antacid use for reflux related to food impaction or with a history of esophageal spasm.
* Patients already tolerating processed/cooked forms of the food (e.g.,baked goods with milk).

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of anaphylaxis in different Oral Immunotherapy protocols | 3 years
  Do participants in the different study arms experience similar rates of anaphylaxis during their participation in the study? Anaphylaxis is defined as an allergic reaction to the food the subject is allergic to, that involves symptoms in two of the following organ systems: skin, respitratory, gastro-enterologic or neurologic.The Consortium for Food Allergy Research (CoFAR) grading scale will be used for assessing severuty of allergic symptoms

SECONDARY OUTCOMES:
Efficacy of different Oral Immunotherapy protocols | 3 years
  Do participants in the three study arms experience similar levels of desensitization to their allergen? This will be assessed by a Double-Blind Placebo Controlled Oral Food Challenge (DBPCFC). Doses of allergen that elicit symptoms strong enough to end the challenge will be compared between the three groups. Symptom severity will be graded using the CoFAR grading scale.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Ben-Shoshan, MD, Principal Investigator — MUHC-RI
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared. All participant data will remain strictly confidential

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT06256146/Prot_SAP_000.pdf